CLINICAL TRIAL: NCT00542997
Title: A Multicentre Study of the Efficacy, Tolerability, Safety, and Pharmacokinetics of Immune Globulin Subcutaneous (Human) IgPro20 in Subjects With Primary Immunodeficiency
Brief Title: Study of Subcutaneous Immune Globulin in Patients Requiring IgG Replacement Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Global Head Clinical R&D, CSL Behring
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1460; ZLB06_001CR (Other: CSL Behring)
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Common Variable Immunodeficiency; X-linked Agammaglobulinemia; Autosomal Recessive Agammaglobulinemia
Keywords: Subcutaneous immune globulin; SCIG
MeSH Terms: conditions — Common Variable Immunodeficiency; Bruton type agammaglobulinemia; Agammaglobulinemia, non-Bruton type | interventions — gamma-Globulins; Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IgPro20 (Experimental)
  Interventions: Biological: Human Normal Immunoglobulin for Subcutaneous Administration (IGSC)

INTERVENTIONS:
Biological: Human Normal Immunoglobulin for Subcutaneous Administration (IGSC) — IgPro20 is a liquid formulation of normal human IgG at a concentration of 20% administered as a SC infusion at weekly intervals. The initial weekly dose was determined based on subjects' previous treatment. Dose adjustments could be performed during the wash-in/wash-out period at the discretion of the investigator.
  Other Names: Hizentra; SCIG

SUMMARY:
The objective of this study is to assess the efficacy, tolerability, safety and pharmacokinetics of IgPro20 in patients with primary humoral immunodeficiency (PID).

DETAILED DESCRIPTION:
This study consisted of a 12-week wash-in/wash-out period followed by a 28-week efficacy period. During the 28-week efficacy period, subjects visited the study site at least every 4 weeks for efficacy and safety evaluations and additionally recorded details regarding IgPro20 dose and certain aspects of efficacy and safety in a diary. Pharmacokinetic (PK) parameters were assessed in a sub-group of subjects during 1 treatment interval at steady-state (Week 28 ± 1).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with primary humoral immunodeficiency, namely with a diagnosis of Common Variable Immunodeficiency (CVID) as defined by the Pan-American Group for Immunodeficiency (PAGID) and European Society for Immunodeficiencies (ESID), X-linked agammaglobulinemia (XLA) as defined by PAGID and ESID, or Autosomal Recessive Agammaglobulinemia
* Chest X-ray or CT scan obtained within 1 year prior to enrolment

Exclusion Criteria:

* Newly diagnosed PID, i.e. subjects who have not previously received immunoglobulin replacement therapy
* Ongoing serious bacterial infection at the time of screening
* Malignancies of lymphoid cells such as lymphocytic leukemia, Non-Hodgkin's lymphoma and immunodeficiency with thymoma
* Allergic or other severe reactions to immunoglobulins or other blood products associated with high anti-IgA

Additional criteria may apply and examination by an investigator is required to determine eligibility.

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Jolles, MD, Principal Investigator — University Hospital of Wales, Cardiff, UK
Locations (19):
- Study site, Paris, France
- Germany (7):
  - Study site, Berlin
  - Study site, Düsseldorf
  - Study site, Freiburg im Breisgau
  - Study site, Hanover
  - Study site, Leipzig
  - Study site, Mainz
  - Study site, Munich
- Study site, Brescia, Italy
- Study site, Warsaw, Poland
- Romania (3):
  - Study site, Bucharest
  - Study site, Cluj-Napoca
  - Study site, Timișoara
- Spain (2):
  - Study site, Barcelona
  - Study site, Seville
- Study site, Gothenburg, Sweden
- Study site, Bern, Switzerland
- United Kingdom (2):
  - Study site, Cardiff
  - Study site, London

REFERENCES:
- [Result] Jolles S, Bernatowska E, de Gracia J, Borte M, Cristea V, Peter HH, Belohradsky BH, Wahn V, Neufang-Huber J, Zenker O, Grimbacher B. Efficacy and safety of Hizentra((R)) in patients with primary immunodeficiency after a dose-equivalent switch from intravenous or subcutaneous replacement therapy. Clin Immunol. 2011 Oct;141(1):90-102. doi: 10.1016/j.clim.2011.06.002. Epub 2011 Jun 12. PMID 21705277
- [Result] Borte M, Pac M, Serban M, Gonzalez-Quevedo T, Grimbacher B, Jolles S, Zenker O, Neufang-Hueber J, Belohradsky B. Efficacy and safety of hizentra(R), a new 20% immunoglobulin preparation for subcutaneous administration, in pediatric patients with primary immunodeficiency. J Clin Immunol. 2011 Oct;31(5):752-61. doi: 10.1007/s10875-011-9557-z. Epub 2011 Jun 15. PMID 21674136

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multinational study enrolled subjects at 15 of the participating study centers in Europe.
Pre-assignment Details: Screening took place 1 to 4 weeks prior to the first IgPro20 infusion.
Groups:
- IgPro20 (All Treated): All subjects receiving at least 1 infusion of IgPro20
Period: Wash in / Wash Out Period
Arm/Group | IgPro20 (All Treated)
Started | 51
Completed | 46
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 3
Period: Efficacy Period
Arm/Group | IgPro20 (All Treated)
Started | 46
Completed | 43
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Groups:
- IgPro20 (All Treated): All subjects enrolled and treated with subcutaneous infusion of IgPro20
Arm/Group | IgPro20 (All Treated)
Number analyzed (Participants) | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 22.6 (16.02)
Age, Customized [Number; unit: Participants]
  2 to < 12 years | 18
  12 to < 16 years | 5
  16 to < 65 years | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 35
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 51
Type of Primary Immunodeficiency [Number; unit: Participants]
  Common variable immunodeficiency (CVID) | 30
  X-linked agammaglobulinemia (XLA) | 20
  Autosomal recessive agammaglobulinemia (ARAG) | 1

OUTCOME MEASURES:

1. Primary Outcome: Total Serum IgG Trough Levels
Description: Total IgG trough levels for IgPro20 treatment at steady state were compared with documented trough level data for IgG treatment received prior to enrolling in the study (either subcutaneous or intravenous IgG). For this purpose, 6 consecutive IgPro20 trough values (obtained prior to infusions 12 to 17) per subject were aggregated to the subject's median value and then median values across subjects were summarised using descriptive statistics. The same procedure was applied to pre-study treatment using the 3 most recent IgG trough values ≥ 5 g/L obtained prior to the first IgPro20 infusion.
Time Frame: Up to 6 months prior to first IgPro20 treatment (Pre-study treatment) and Week 12 to 17 (IgPro20 treatment)
Population: Intention-to-treat (ITT) population analysis. The ITT population included all subjects who were treated with IgPro20 during the efficacy period (starting with Week 12). For 2 subjects in the ITT population, the pre-study treatment IgG trough levels were not available.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- IgPro20: Subjects enrolled and treated with subcutaneous infusion of IgPro20 during the Efficacy Period (Infusions 12 to 17)
- Pre-study IgG Treatment: Enrolled subjects with at least 3 documented IgG trough values ≥ 5 g/L during up to 6 months of intravenous (IGIV) or subcutaneous (IGSC) replacement therapy prior to receiving IgPro20 study treatment.
Arm/Group | IgPro20 | Pre-study IgG Treatment
Number analyzed (Participants) | 46 | 44
g/L | 8.10 (1.44) | 7.49 (1.57)

2. Secondary Outcome: Annual Rate of Clinically Documented Serious Bacterial Infections (ITT Population)
Description: Serious bacterial infections (SBIs) included bacterial pneumonia, bacteraemia/septicaemia, osteomyelitis/septic arthritis, bacterial meningitis, and visceral abscess. Diagnosis of the SBIs was based on the presence of predefined clinical signs and symptoms as well as on laboratory parameters.
  The annual rate was calculated based on the total number of SBIs and the total number of study days during the efficacy period for all subjects in the ITT population and adjusted to 365 days.
Time Frame: Efficacy period: week 12 to week 40 after study start or to the completion visit
Population: Intention-to-treat (ITT) population analysis. The ITT population included all subjects who were treated with IgPro20 during the efficacy period (starting with Week 12).
Measure: Number; unit: SBIs/subject/year
Units Other Than Participants: Subject Days
Groups:
- IgPro20: Subjects enrolled and treated with subcutaneous infusion of IgPro20
Arm/Group | IgPro20
Number analyzed (Participants) | 46
Number analyzed (Subject Days) | 8745
SBIs/subject/year | 0

3. Secondary Outcome: Annual Rate of Clinically Documented Serious Bacterial Infections (PPE Population)
Description: Serious bacterial infections (SBIs) included bacterial pneumonia, bacteraemia/septicaemia, osteomyelitis/septic arthritis, bacterial meningitis, and visceral abscess. Diagnosis of the SBIs was based on the presence of predefined clinical signs and symptoms as well as on laboratory parameters.
  The annual rate was calculated based on the total number of SBIs and the total number of study days during the efficacy period for all subjects in the PPE population and adjusted to 365 days.
Time Frame: Efficacy period: week 12 to week 40 after study start or to the completion visit
Population: Per Protocol Efficacy (PPE) population analysis. The PPE population included all subjects who completed the 28-week efficacy period according to protocol.
Measure: Number; unit: SBIs/subject/year
Units Other Than Participants: Subject Days
Arm/Group | IgPro20
Number analyzed (Participants) | 34
Number analyzed (Subject Days) | 6729
SBIs/subject/year | 0

4. Secondary Outcome: Annual Rate of Infection Episodes
Description: The annual rate of episodes was calculated based on the total number of any infection type and the total number of study days during the efficacy period for all subjects in the ITT population and adjusted to 365 days.
Time Frame: Efficacy period: week 12 to week 40 after study start or to the completion visit
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: episodes/subject/year
Units Other Than Participants: Subject Days
Arm/Group | IgPro20
Number analyzed (Participants) | 46
Number analyzed (Subject Days) | 8745
episodes/subject/year | 5.18 [4.31 to 6.17]

5. Secondary Outcome: Annual Rate of Days Out of Work / School / Kindergarten / Day Care or Unable to Perform Normal Activities Due to Infections
Description: The annual rate was calculated based on the total number of days out of work/school/kindergarten/day care or unable to perform normal activities due to infections in the efficacy period divided by the total number of days in the efficacy period for all subjects and adjusted to 365 days.
Time Frame: Efficacy period: week 12 to week 40 after study start or to the completion visit
Population: as for outcome 2
Measure: Number; unit: days/subject/year
Units Other Than Participants: Subject Days
Arm/Group | IgPro20
Number analyzed (Participants) | 46
Number analyzed (Subject Days) | 9033
days/subject/year | 8.00

6. Secondary Outcome: Annual Rate of the Number of Days of Hospitalization Due to Infections
Description: The annual rate was calculated based on the total number of days of hospitalization due to infections in the efficacy period divided by the total number of days in the efficacy period for all subjects and adjusted to 365 days.
Time Frame: Efficacy period: week 12 to week 40 after study start or to the completion visit
Population: ITT population analysis.
  The intention-to-treat (ITT) data set comprises all subjects treated with the study drug during the efficacy period (week 13 to week 40 after study start or to the completion visit).
Measure: Number; unit: days/subject/year
Units Other Than Participants: Subject Days
Arm/Group | IgPro20
Number analyzed (Participants) | 46
Number analyzed (Subject Days) | 9033
days/subject/year | 3.48

7. Secondary Outcome: Annual Rate of Antibiotic Use for Infection Prophylaxis and Treatment
Description: The annual rate was calculated based on the total number of days of antibiotic use in the efficacy period divided by the total number of days in the efficacy period for all subjects and adjusted to 365 days.
Time Frame: Efficacy period: week 12 to week 40 after study start or to the completion visit
Population: as for outcome 6
Measure: Number; unit: days/subject/year
Units Other Than Participants: Subject Days
Arm/Group | IgPro20
Number analyzed (Participants) | 46
Number analyzed (Subject Days) | 8745
days/subject/year | 72.75

8. Other Pre Specified Outcome: Maximum Concentration (Cmax) of Total Serum IgG
Time Frame: Week 28 (±1week)
Population: Per Protocol Pharmacokinetic (PPK) population analysis. A total of 24 of the 51 enrolled subjects were included in a pharmacokinetic (PK) sub-study. 23 subjects completed the PK sub-study per protocol and were included in the PPK analysis population.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- IgPro20 (PK Substudy): Subjects enrolled and treated with subcutaneous infusion of IgPro20 participating in the pharmacokinetic sub-study
Arm/Group | IgPro20 (PK Substudy)
Number analyzed (Participants) | 23
g/L | 8.26 (1.25)

9. Other Pre Specified Outcome: Timepoint of Maximum Concentration (Tmax) of Total Serum IgG
Time Frame: Week 28 (±1week)
Population: as for outcome 8
Measure: Median (Full Range); unit: day
Arm/Group | IgPro20 (PK Substudy)
Number analyzed (Participants) | 23
day | 2.06 [0.94 to 6.92]

10. Other Pre Specified Outcome: Area Under the Concentration-Time Curve (AUC_last) of Total Serum IgG
Description: AUC_last = Area under the concentration-time curve until last measured concentration.
Time Frame: Week 28 (±1week)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day x g/L
Arm/Group | IgPro20 (PK Substudy)
Number analyzed (Participants) | 23
day x g/L | 53.70 (9.16)

11. Other Pre Specified Outcome: Area Under the Concentration-Time Curve (AUCτ) of Total Serum IgG
Description: AUCτ = Area under the concentration-time curve during regular dosing interval;
Time Frame: Week 28 (±1week)
Population: Per Protocol Pharmacokinetic (PPK) population analysis. A total of 24 of the 51 enrolled subjects were included in a pharmacokinetic (PK) sub-study. 23 subjects completed the PK sub-study per protocol and were included in the PPK analysis population. 7 subjects were missing data for AUCτ.
Measure: Mean (Standard Deviation); unit: day x g/L
Arm/Group | IgPro20 (PK Substudy)
Number analyzed (Participants) | 16
day x g/L | 53.61 (9.98)

ADVERSE EVENTS:
Time Frame: The observation period for adverse events was from the time the subjects had given informed consent until they had the final examination (completion visit up to 40 weeks) or extended when serious adverse events were reported.
Description: A total of 1831 infusions of IgPro20 were administered to 51 subjects during the course of the study.
Arm/Group | IgPro20 (All Treated)
Serious Adverse Events (participants affected / at risk) | 5/51
Other Adverse Events (participants affected / at risk) | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (All Treated) (N=51)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2)
Pyrexia (General disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro20 (All Treated) (N=51)
Bronchitis (Infections and infestations) | 16 (26)
Pyrexia (General disorders) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (26)
Headache (Nervous system disorders) | 13 (54)
Nasopharyngitis (Infections and infestations) | 12 (20)
Upper respiratory tract infection (Infections and infestations) | 12 (17)
Diarrhoea (Gastrointestinal disorders) | 10 (16)
Injection site reaction (General disorders) | 9 (16)
Sinusitis (Infections and infestations) | 7 (11)
Injection site pain (General disorders) | 6 (8)
Infusion site pain (General disorders) | 5 (10)
Injection site pruritus (General disorders) | 5 (17)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Injection site swelling (General disorders) | 4 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (14)
Respiratory tract infection (Infections and infestations) | 4 (5)
Vomiting (Gastrointestinal disorders) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4)
Acute sinusitis (Infections and infestations) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Conjunctivitis (Eye disorders) | 3 (6)
Erythema (Skin and subcutaneous tissue disorders) | 3 (5)
Fatigue (General disorders) | 3 (6)
Gastroenteritis (Infections and infestations) | 3 (3)
Infusion site haematoma (General disorders) | 3 (3)
Injection site erythema (General disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Oral herpes (Infections and infestations) | 3 (3)
Rhinitis (Infections and infestations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to public release. The sponsor may request any changes necessary to prevent forfeiture of patent rights to data not in the public domain. For a multi-center study, the investigator must wait (i) at least 1 year after the study is completed at all sites or (ii) until notified by the sponsor that no multi-center publication is planned before seeking publication review.